CLINICAL TRIAL: NCT00504322
Title: Phase II, Randomized, Double-blinded, Placebo-Control, Toxicity/Efficacy Study on the Transfer of Adenovirus With the CD40 Ligand Gene (AdcuCD40L) to Patients With Stage I, II or III Esophageal Carcinoma
Brief Title: Efficacy Study on the Transfer of Adenovirus With the CD40 Ligand Gene (AdcuCD40L) to Patients With Esophageal Carcinoma
Acronym: cd40
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding available.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0502007770
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): The placebo will be the salt water-sugar solution used as a vehicle for the vector.
  Interventions: Genetic: Placebo
- AdcuCD40L (Active Comparator): Using Weill-IRB protocol #0011004683 dose escalation study to determine the highest non-toxic dose of the AdcuCD40L vector, this dose (likely 10^11 particle units) will be used for all individuals enrolled in this efficacy study. Since there is no evidence that delay of surgery for solid tumors for 15 days following diagnosis alters the prognosis, surgery for removal of the primary tumor will be carried out at either 5 or 15 days after administration of the vector (n= 12/group, including n=6 receiving the AdcuCD40L vector, and n=6 receiving placebo). This will permit assessment of the resulting data (in a randomized, blinded fashion) and the biologic responses to the AdCUCD40L vector over time.
  Interventions: Genetic: AdcuCD40L

INTERVENTIONS:
Genetic: AdcuCD40L — Using Weill-IRB protocol #0011004683 dose escalation study to determine the highest non-toxic dose of the AdcuCD40L vector, this dose (likely 10^11 particle units) will be used for all individuals enrolled in this efficacy study. Since there is no evidence that delay of surgery for solid tumors for 15 days following diagnosis alters the prognosis, surgery for removal of the primary tumor will be carried out at either 5 or 15 days after administration of the vector (n= 12/group, including n=6 receiving the AdcuCD40L vector, and n=6 receiving placebo). This will permit assessment of the resulting data (in a randomized, blinded fashion) and the biologic responses to the AdCUCD40L vector over time.
  Other Names: Active Comparator
  Arms: AdcuCD40L
Genetic: Placebo — The placebo will be the salt water-sugar solution used as a vehicle for the vector.
  Other Names: salt water-sugar solution
  Arms: placebo

SUMMARY:
This study is a randomized, double-blinded assessment of biologic efficacy of AdcuCD40L. The individuals enrolled in this study will be individuals with biopsy proven resectable esophageal carcinoma. The dose of the AdcuCD40L vector (administered endoscopically directly to the tumor) will be the highest tolerable dose (most likely 10^11 particle units) determined from Weill-IRB protocol #0011004683 dose escalation study.

DETAILED DESCRIPTION:
This study is designed to add to the safety profile data as well as assessing biologic efficacy parameters. It will include 24 individuals with biopsy proven, resectable, stage I-III esophageal cancer. Because there may be immune responses attributable to the gene therapy vector itself, independent of the CD40L transgene, this part of the study is designed in a randomized, blinded fashion to compare intratumoral administration of the AdcuCD40L vector compared to a placebo. Because there are likely differences over time in the pattern of the biologic response to the expression of CD40L in the tumor (including activation and trafficking of DC, and recruitment and activation of immune cells), this study will include 2 "time" cohorts (based on the time between administration of the AdcuCD40L vector and the time of surgery to remove the tumor). Using Weill-IRB protocol #0011004683 dose escalation study to determine the highest non-toxic dose of the AdcuCD40L vector, this dose (likely 10^11 particle units) will be used for all individuals enrolled in this efficacy study. The placebo will be the salt water-sugar solution used as a vehicle for the vector. Since there is no evidence that delay of surgery for solid tumors for 15 days following diagnosis alters the prognosis, surgery for removal of the primary tumor will be carried out at either 5 or 15 days after administration of the vector (n= 12/group, including n=6 receiving the AdcuCD40L vector, and n=6 receiving placebo). This will permit assessment of the resulting data (in a randomized, blinded fashion) and the biologic responses to the AdCUCD40L vector over time. In addition to safety/toxicity parameters, the primary tumor, regional and distant nodes removed at the time of surgery, and peripheral blood will be assessed for biologic parameters relevant to responses to the AdcuCD40L vector.

ELIGIBILITY:
Inclusion Criteria:

* Must be capable of providing informed consent
* Males and females, age 18 to 75 years
* Hematocrit > 30%
* WBC < 10,000
* Normal prothrombin, partial thromboplastin time; platelet count > 100,000
* Normal liver-related serum parameters
* Blood urea nitrogen < 60 mg/dL, creatinine < 2.5 mg/dl
* No evidence of active infection of any type, including with adenovirus, hepatitis virus (A, B or C), or human immunodeficiency virus
* No evidence of central nervous system, major psychiatric, musculoskeletal, or immune disorder
* No allergy to the vehicle used to suspend the virus or contrast materials used in radiographic procedures
* Fertile or infertile individuals; it will be recommended that fertile individuals utilize barrier birth control measures to prevent pregnancy during and for 1 month following the administration of the vector
* Biopsy proven esophageal cancer; clinically stage I-III, deemed resectable by the patient's surgeon. No history of neoadjuvant chemotherapy or chemoradiotherapy. Distant metastases are to be ruled out at the discretion of the physician treating the patient according to standards of care
* Individuals not receiving experimental medications or participating in another experimental protocol for at least 4 weeks prior to entry to the study
* The study individual must be able to undergo the procedures in the protocol
* Willingness to participate in the study

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria will be unable to participate in the protocol
* Individuals in whom participation in the study would compromise the normal care and expected progression of their disease
* Individuals receiving corticosteroids or other immunosuppressive medications; previous splenectomy or radiation to the spleen; autoimmune disease
* Recent (less than 6 week) cerebral vascular accident
* Recent (less than 6 week) transmural myocardial infarction
* Evidence of infection defined by elevated white blood cell count, temperature > 38.5oC or infiltrate on chest x-ray
* Cervical esophageal cancer
* Gastric cancer (tumor more than 50% in the stomach as determined by endoscopy)
* Pathology other than squamous cell or adenocarcinoma
* Malignant ventricular arrhythmia
* Pregnancy
* Immunodeficiency disease, including evidence of HIV infection
* Current alcohol or drug abuse
* Esophageal tumor too small for adequate tissue harvest (determined during esophagoscopy at the time of vector or placebo injection)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Expression of CD40L and cytokines | 5-15 days

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Crystal, MD, Principal Investigator — Department of Genetic Medicine

IPD SHARING:
Plan to Share IPD: Undecided